CLINICAL TRIAL: NCT02648516
Title: Safety and Efficacy of Allogenic Adoptive Immune Therapy for Immune Reconstitution Failure in Chronic HIV-1 Infected Patients
Brief Title: Safety and Efficacy of Allogenic Adoptive Immune Therapy for Immune Reconstitution in Chronic HIV-1 Infected Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Beijing302-010
Record Dates: First submitted 2015-09-08; First posted 2016-01-07 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-05

CONDITIONS: Human Immunodeficiency Virus; Disorder of Immune Reconstitution
Keywords: Immune Reconstitution; Allogenic HLA-Mismatched Mononuclear Cells Transplantation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Congresses as Topic; AaIT neurotoxin, Androctonus australis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Conventional plus AAIT (Experimental): Participants will receive ART plus a dose of allogenic adoptive immune transfusion (3 times of MNCs transfusions) from day 0 through the week 2 study visit.
  Interventions: Combination Product: Conventional plus AAIT

INTERVENTIONS:
Combination Product: Conventional plus AAIT — Participants will receive ART and taken i.v., at a dose of 2-3*10E8 MNCs/kg body at baseline, week 1 and 2.
  Other Names: Conventional plus allogenic adoptive immune treatment

SUMMARY:
Combination antiretroviral therapy (ART) effectively suppresses viral replication, leading to a significant immune recovery and a dramatic reduction in the incidence of AIDS-defining events. However, approximately 20% of individuals who exhibit stable viral suppression by ART, but fail to achieve sufficient immune reconstitution and are considered immune nonresponders (INRs). These INRs often experience an increased risk of opportunistic infections and shorter life expectancy compared with matched immune responders.Therefore, efficiently treating these immune nonresponders has become one of the most difficult challenges in the clinic.

DETAILED DESCRIPTION:
There is not a consensus definition of immunologic nonresponder individuals. In this study, we described patients whose cluster of differentiation 4（CD4)+ T-cell count remained below 200 cells/ul after 2 years of effective antiviral as immunologic nonresponders, in which viroimmunological dissociation implies a greater risk of AIDS related and non-AIDS-related illnesses. Immune-based therapy such as interleukin (IL)-2 and IL-7 have been shown to increase CD4 T-cell counts but yielded no clinical benefit in a large randomized study. We have reported that umbilical cord Tissue Mesenchymal Stem Cells (UC-MSC) treatment is safe and can significantly decrease systemic immune overactivation and improve immune reconstitution in INR patients. Meanwhile, we did not find that there was a significantly transitory increase in peripheral CD4 T-cell counts within 1-2 weeks since the onset of each MSC infusion. More important, umbilical cord-MSCs were found to be with a potential to produce IL-7 and T-cell growth factor transforming growth factor (TGF)-β in vitro and in vivo and preferentially expand CD4 T-cell response in the recipients. Therefore, development of novel interventions to reduce immune overactivation/inflammation and enhance immune reconstitution in INRs is a high priority.

Granulocyte colony-stimulating factor (G-CSF)-mobilized donor peripheral blood mononuclear cells (MNCs) are a heterogeneous population of immune cells that have a potential role in immunomodulation and hemopoiesis. Here, we hypothesized that human leukocyte antigen (HLA)-mismatched MNCs transfusion can be used to comprehensively restore or boost the host holistic immune system for INR patients, to the degree similar as immune responders.

The purpose of this study is to investigate the safety and initial efficacy of allogeneic adoptive immune therapy (AAIT) for INR patients. 20 INR patients received i.v. transfusion one round (3 times) of 2.0-3.0*10E8 cells/kg of MNCs as the treated group. All of them received the conventional treatment for AIDS. The CD4 T cell numbers, HIV reservoir, side effects, symptom improvement, control of opportunistic infections and will be evaluated during the 96-week follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Immune non-responders with chronic HIV-1 infection
2. Antiretroviral therapy (ART) for at least 24 months prior to study entry and continue within the 24 months after study entry
3. CD4 count less than or equal to 200 cells/mm3 continuously and more than 50 cells/mm3 before entry and at screening, obtained within 30 days prior to study entry
4. Viral load less than or equal to 50 copies/mL obtained within 12 months prior to study entry
5. Certain specified laboratory values obtained within 30 days prior to study entry. More information on this criterion can be found in the study protocol
6. Documentation that pre-entry specimen for the primary immune activation endpoint responses has been obtained
7. No history of Centers for Disease Control and Prevention (CDC) category C AIDS-related opportunistic infections
8. Karnofsky performance score greater than or equal to 70 within 30 days prior to study entry
9. Ability and willingness to provide informed consent

Exclusion Criteria:

1. Coinfection with other virus, including serum hepatitis C virus RNA positive, or one of followings are positive in anti-hepatitis A virus/anti-HDV/anti-hepatitis delta virus plus alanine aminotransferase (ALT) more than 80 IU/L
2. History of combination with other severe diseases including renal, circulatory, respiratory, digestive, endocrine, neural and immunological diseases and tumors
3. White blood cell (WBC) <2.5*10E9/L, platlet counts <50*10E9/L, Hb <80g/L, lactate >2 mmol/L
4. Allergic constitution
5. Pregnancy or lactation
6. Accepting other immunomodulatory drugs within 6 months prior screening
7. Drug addiction
8. Other conditions possibly influencing the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The changes of CD4 T cell counts | At Baseline and week 1, 2, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96
  marker for host immunity

SECONDARY OUTCOMES:
The changes of HIV-1 DNA | At Baseline and up to week 96
  marker for HIV-1 reservoir
The ratio of CD4 and CD8 T cells | At Baseline and week 1, 2, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96
  marker for host immunity
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | At Baseline and up to week 96
  marker for safety

CONTACTS AND LOCATIONS:
Overall Officials: Wang Fu-Sheng, Principal Investigator — Beijing 302 Hospital
Locations (1):
- Beijing 302 hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Z, Fu J, Xu X, Wang S, Xu R, Zhao M, Nie W, Wang X, Zhang J, Li T, Su L, Wang FS. Safety and immunological responses to human mesenchymal stem cell therapy in difficult-to-treat HIV-1-infected patients. AIDS. 2013 May 15;27(8):1283-93. doi: 10.1097/QAD.0b013e32835fab77. PMID 23925377
- [Background] Hutter G. Stem cell transplantation in strategies for curing HIV/AIDS. AIDS Res Ther. 2016 Sep 13;13(1):31. doi: 10.1186/s12981-016-0114-y. eCollection 2016. PMID 27625700
- [Background] Corbeau P, Reynes J. Immune reconstitution under antiretroviral therapy: the new challenge in HIV-1 infection. Blood. 2011 May 26;117(21):5582-90. doi: 10.1182/blood-2010-12-322453. Epub 2011 Mar 14. PMID 21403129